CLINICAL TRIAL: NCT03254576
Title: Cue-Reward Learning and Weight Gain in Youth
Acronym: ChildLearn
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kerri Boutelle, Professor, University of California, San Diego
Other Study IDs: 161468; R01DK111106 (NIH)
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Body Mass Index; Weight; Brain imaging; Child; Learning
MeSH Terms: conditions — Overweight; Obesity; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children at high-risk for obesity: Healthy-weight children (5th-75thBMI%) with two overweight/obese parents (BMI>25)
  Interventions: Other: Functional MRI
- Children at low-risk for obesity: Healthy-weight children (5th-75thBMI%) with two healthy-weight parents (BMI = 18-24.9)
  Interventions: Other: Functional MRI

INTERVENTIONS:
Other: Functional MRI

SUMMARY:
The objective of the study is to compare children at low risk for obesity (two healthy weight parents) to children at high risk for obesity (two overweight parents) in their response rate to food taste and in their rate of learning using fMRI.

DETAILED DESCRIPTION:
The primary aim of this project is to conduct an adequately powered study that compares children at low risk for obesity to children at high risk for obesity on their brain responses to food tastes during a pavlovian learning task. Seven assessment visits will be conducted at three separate time points; baseline, 1-year follow up, and 2-year follow up. Assessments will include anthropometry, interviews, computer tasks, questionnaires, and an fMRI scan. This program of research tests a novel hypothesis regarding overeating and the development of obesity in children, and could provide critical data on individual vulnerabilities to overeating for further research. Furthermore, this study could provide mechanisms for intervention with regards to cue-reward learning in children, to ultimately prevent obesity in youth.

ELIGIBILITY:
Inclusion Criteria:

* Healthy weight children between the ages of 8 and 11 Years
* BMI 5-75th percentile
* Child must be right-handed
* Child must be willing to participate in an fMRI scan
* Either two biological parents who are overweight/obese or no biological parents that are overweight/obese
* One biological parent willing to bring child to assessment visits
* Child and participating parent Fluent in English for speaking, reading, and writing
* Child must like cheese pizza and chocolate milkshake

Exclusion Criteria:

* Child overweight (BMI≥85th percentile)
* Child diagnoses of a serious chronic physical disease (e.g., diabetes) for which physician supervision of diet and exercise prescription are needed
* Child who is taking medications that may impact brain responses (can take kids who are stable on meds)
* Child with MRI contraindications (presence of metallic foreign object or device in body, piercings that cannot be removed, tattooed permanent makeup that contain metal, braces, head trauma, claustrophobia, use of Bigen permanent hair dye)
* Child with an active eating disorder (reported on EDE interview) or with first degree relative with Anorexia Nervosa or Bulimia Nervosa
* Cognitive impairment or disability determined through parent and child self-report measures, and parent reported child individual education plan
* Vision problems uncorrectable with lenses
* Food allergies related to cheese pizza, chocolate milkshake, or the snack foods used in the study
* Menarche in female participants at time of enrollment
* Children scoring within the midpubertal range or higher based on the Pubertal Development Scale

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy-weight children (5-75thBMI%) between the ages of 8 and 11 years old with either two over-weight parents (BMI>25) or two healthy-weight parents (BMI = 18-24.9)
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Cue-reward learning | Baseline only
  Whether rate of the shift in BOLD response from food cue to neutral cue is different between high and low-risk children
Reward Sensitivity | Baseline only
  Whether the BOLD response to food cue differs between high and low-risk children
Weight gain | Change from baseline at an average of 12 months and 24 months
  Whether rate of cue reward and reward sensitivity predict weight gain

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, Ph.D., Principal Investigator — UCSD
Locations (1):
- UCSD Center for Healthy Eating and Activity Research (CHEAR), La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boutelle KN, Wierenga CE, Bischoff-Grethe A, Melrose AJ, Grenesko-Stevens E, Paulus MP, Kaye WH. Increased brain response to appetitive tastes in the insula and amygdala in obese compared with healthy weight children when sated. Int J Obes (Lond). 2015 Apr;39(4):620-8. doi: 10.1038/ijo.2014.206. Epub 2014 Dec 11. PMID 25582522
- [Background] Mestre ZL, Bischoff-Grethe A, Eichen DM, Wierenga CE, Strong D, Boutelle KN. Hippocampal atrophy and altered brain responses to pleasant tastes among obese compared with healthy weight children. Int J Obes (Lond). 2017 Oct;41(10):1496-1502. doi: 10.1038/ijo.2017.130. Epub 2017 Jun 2. PMID 28572588